CLINICAL TRIAL: NCT00765622
Title: Assessment of Pelvic Floor Function in Women With Urinary Incontinence
Brief Title: Assessment of Pelvic Floor Function in Elderly
Status: Completed | Type: Observational
Sponsor: Catholic University of Brasília (Other)
Responsible Party: Ricardo Jacó de Oliveira, Catholic University of Brasilia
Other Study IDs: ucb123cestari
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-08

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; pelvic floor; functional evaluation
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Women
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- G2: G2 = control group (no incontinence)
- G1: G1 = urinary incontinence

SUMMARY:
The purpose of this study is to demonstrate the importance of functional assessment of the pelvic floor (AFA) in older women, as prognostic factor for Urinary Incontinence (UI).

DETAILED DESCRIPTION:
Incontinence elderly assessment

ELIGIBILITY:
Inclusion Criteria:

* Elderly women
* Urinary incontinence

Exclusion Criteria:

* Cesarean surgery

Ages: 58 Years to 87 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: elderly women
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
All patients were submitted for review physiotherapeutic through palpation bidigital and quantification of contraction pelvic, was performed using a my feedback of pressure | Only one measure at the begging of the study

CONTACTS AND LOCATIONS:
Overall Officials: Claudia EC Souza, Ms, Principal Investigator — Catholic University of brasilia
Locations (1):
- UC, Brasília, Federal District, Brazil